CLINICAL TRIAL: NCT04038749
Title: Satisfaction of Patients With the Chosen Method of Inhibition of Lactation: With the Use of Drugs Lowering the Level of Prolactin or Without the Use of Pharmacological Agents in Postnatal Period, Taking Into Account Individual Conditions
Brief Title: Satisfaction of Patients With the Chosen Method of Inhibition of Lactation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Żelazna Medical Centre, LLC (Other)
Responsible Party: Principal Investigator, Alicja Misztal, Investigator, Żelazna Medical Centre, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23/2019
Record Dates: First submitted 2019-07-17; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Lactation Suppressed
MeSH Terms: interventions — Bromocriptine; Cabergoline; Natural Family Planning Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pharmaceutical method- Bromocriptine (Experimental)
  Interventions: Drug: Bromocriptine; Other: Natural methods
- Pharmaceutical method- Cabergoline (Experimental)
  Interventions: Drug: Cabergoline; Other: Natural methods
- Without medications that inhibit lactation (Other)
  Interventions: Other: Natural methods

INTERVENTIONS:
Drug: Bromocriptine — Bromocriptine - on the first day of treatment (1,25 mg) with morning and evening meal and then 2,5 mg dose twice a day for two weeks (14 days)
  Other Names: Bromergon
  Arms: Pharmaceutical method- Bromocriptine
Drug: Cabergoline — Cabergoline - one dose (1 mg) on the first day after childbirth or 0.25 mg dose every 12 hours for 2 days
  Other Names: Dostinex
  Arms: Pharmaceutical method- Cabergoline
Other: Natural methods — milk expression, cold compress, cabbage leaf compresses, mild painkiller- e.g. ibuprofen, supportive bra, sage tea.

SUMMARY:
The aim of the study is to improve the standard of care in case of the inhibition of lactation.

The participant qualified for the study will answer the questions contained in the survey. The patient will have her breast palpated and then will be instructed on the possible options for the inhibition of lactation. The participant, who decides to inhibit lactation with medications, will be consulted by a doctor.

Each patient will receive information of the possible ways to relieve the symptoms of overfilled breast and be able to contact with lactation consultant. The participant will also receive a card to assess the severity of symptoms in the following days. The investigators will call the patient between the third and fifth day by phone.

Once again, after 2 weeks from the beginning of the inhibition of lactation in order to ask questions contained in the survey (the course of the process, problems that occurred and the level of satisfaction with the chosen method).

ELIGIBILITY:
Inclusion Criteria:

* Mother during the period of six weeks after childbirth
* Decision to inhibit lactation
* Patient's age at the time of enrollment (at least 18 years old)

Exclusion Criteria:

* Less than 18 years of age
* Lack of patient's consent
* To the pharmacotherapy group- contraindications for the use of the medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | from the 1st day of the inhibition of lactation to 14th day of process
  Pain assesment by Visual Analogue Scale (VAS scale), range 0-10, higher numbers represents worse outcome.
Evaluation of breast status | from the 1st day of the inhibition of lactation to 14th day of process
  Daily evaluation of breast status. Are they: heavy, full, swollen (engorged), warmed up, hard, irregular, leaking. Gradations of symptoms intensity by using (+) and (-) where:
  * "-" - means not at all
  * "+" - means a little
  * "++" - means a lot
  * "+++" - means very (highest level)
Symptoms in association with the ingestion of medicines that inhibit lactation. | from the 1st day of the inhibition of lactation to 14th day of process
  * headache
  * constipation
  * stomach pain
  * general weakness
  * somnolence
  * vomiting
  * dizziness
  * nausea
  * other
  Symptoms that occurred are marked with a "+".
Breast palpation | 1st day of including in the study
  • Size (each one separately; left and right breast)
  * hypoplastic
  * small
  * average
  * big
  The correct answer is marked with a "+".
  • Anomalies (each one separately; left and right breast)
  * no change
  * swollen
  * redness
  * warming
  * achiness
  * scars
  The correct answer is marked with a "+".
Survey: 1st day of including in the study | 1st day of including in the study
  Questions about:
  * parturition,
  * previous lactations,
  * cause of lactation suppression,
  * factors which may impair lactation,
  * contraindications to medications that suppress lactation,
  * current lactation,
  * the way to suppress lactation.

SECONDARY OUTCOMES:
Survey: 3rd-5th day of lactation suppression | 3rd-5th day of lactation suppression
  Question about:
  • ailments, problems and extra methods of relief of symptoms
Survey: 14th-16th day of lactation suppression | 14th-16th day of lactation suppression
  Questions about:
  * specific ailments and problems during the inhibition of lactation process (such as. pain, feeling of heaviness, temperature, low-grade fever/higher fever, stasis, mastitis, breast abscess, side effects caused by medications)
  * applied methods to ease ailments: (milk expression, cold compress, cabbage leaf compresses, mild painkiller- e.g. ibuprofen, supportive bra, sage tea).
  * assessment whether the decision on how to inhibit lactation was right

CONTACTS AND LOCATIONS:
Overall Officials: Dorota Sys, PhD, Study Chair — Centre of Postgraduate Medical Education
Locations (1):
- Żelazna Medical Centre, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No